CLINICAL TRIAL: NCT05800587
Title: Phase II Study of Dose Attenuated Chemotherapy in Patients With Lung Cancer and Age > 70 and/or Comorbidities
Brief Title: Dose Attenuated Chemotherapy in Compromised Patients With Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-1052; TH-214 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2023-03-24; First posted 2023-04-05 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer; Small-cell Lung Cancer; Non Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Pemetrexed; Paclitaxel; Taxes; Docetaxel; Gemcitabine; Etoposide; Irinotecan; Topotecan; PM 01183

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Platinum doublet plus immunotherapy (IO) (Experimental)
  Interventions: Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Nab paclitaxel; Drug: Docetaxel; Drug: Gemcitabine; Drug: Etoposide; Drug: Irinotecan; Drug: Topotecan; Drug: Lurbinectedin
- Platinum doublet with or without a VEGFi (Experimental)
  Interventions: Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Nab paclitaxel; Drug: Docetaxel; Drug: Gemcitabine; Drug: Etoposide; Drug: Irinotecan; Drug: Topotecan; Drug: Lurbinectedin
- Single agent chemotherapy with or without a VEGFi (Experimental)
  Interventions: Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Nab paclitaxel; Drug: Docetaxel; Drug: Gemcitabine; Drug: Etoposide; Drug: Irinotecan; Drug: Topotecan; Drug: Lurbinectedin

INTERVENTIONS:
Drug: Carboplatin — Standard of care chemotherapy regimen
Drug: Pemetrexed — Standard of care chemotherapy regimen
Drug: Paclitaxel — Standard of care chemotherapy regimen
Drug: Nab paclitaxel — Standard of care chemotherapy regimen
Drug: Docetaxel — Standard of care chemotherapy regimen
Drug: Gemcitabine — Standard of care chemotherapy regimen
Drug: Etoposide — Standard of care chemotherapy regimen
Drug: Irinotecan — Standard of care chemotherapy regimen
Drug: Topotecan — Standard of care chemotherapy regimen
Drug: Lurbinectedin — Standard of care chemotherapy regimen

SUMMARY:
This is an open-label, non-randomized, single-center, phase II study to evaluate the efficacy, toxicity and, tolerability of pre-specified dose attenuated chemotherapy regimens in lung cancer patients with comorbidities.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, single-center, phase II study to evaluate the efficacy, toxicity and, tolerability of pre-specified dose attenuated chemotherapy regimens in lung cancer patients with comorbidities. The investigator will indicate the rationale(s) for dose modification based on the subgroups of patients listed in the protocol. Patients may fit into multiple subgroups and this is accounted for in the prospectively defined dose reduction level as listed in the protocol. Prespecified doses by chemotherapeutic agent and dose level adjustment based on patient characteristics and comorbidities are listed in the protocol. Analyses will be stratified by treatment group 1-3 based on the treating physician's selected therapy.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed stage IV (AJCC version 8) lung cancer (small cell or non-small cell). Patients with stage III disease who are not felt to be candidates for definitive therapy are also eligible.
* Must fit into at least one of the subgroups of patients as defined in section 3.3.
* Patients must have planned therapy with a regimen that includes at least one cytotoxic agent as listed in Table 1 (e.g. platinum, taxane, anti-metabolite, vinca alkaloid, podophylotoxin, camptothecin, lurbinectidin etc).
* Must have measurable disease as per RECIST criteria 1.1.
* History of treated or untreated asymptomatic CNS metastases are eligible, provided they meet all of the following criteria:
* No ongoing requirement for corticosteroids as therapy for CNS disease
* No stereotactic radiation or whole-brain radiation within 7 days prior to treatment initiation
* Stable doses of anti-seizure medications are allowed if CNS disease has been treated and is stable. Treatment of CNS disease can include surgery, radiation or response to prior systemic therapy.
* May have received prior therapy for lung cancer. There is no limit on the number of prior therapies.
* Age > 18 years
* ECOG performance status of 0-3
* Ability to understand and willingness to sign a written informed and HIPAA consent documents.
* Females of child-bearing potential must be willing to use an effective method of contraception for the course of the study through at least 6 months after the last dose of study medication.
* Patients with known HIV infection and are receiving combination antiretroviral therapy with a viral load <400 copies per mL at screening or CD4+ T-cell count > 350 cell per μL at screening and no history of AIDS-defining opportunistic infection < 12 months before first dose of study drug are eligible.
* Males who are fertile and who have partners who are Women of Child-bearing Potential (WOCBP) must agree to use effective method(s) of contraception as outlined in section 4.4 from the start of trial treatment, for the course of the study and 6 months after the last dose of study treatment.

Exclusion Criteria:

* Patients receiving only a targeted agent (e.g. TKI, sotorasib etc.) or immunotherapy without a cytotoxic agent.
* Patients currently receiving investigational agents for cancer.
* Patients with ECOG PS 3 and hepatic or renal dysfunction.
* Clinical signs of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding.
* Undergone major surgery within 28 days prior to first dose of study treatment. The patient has elective or planned major surgery to be performed during the course of the clinical trial.
* Have not recovered from adverse events due to anticancer agents administered previously except neuropathy, alopecia or endocrinopathies that can be treated with replacement therapy. Physician's discretion is allowed to decide which unresolved adverse events from previous therapy prohibit patient participation in this study.
* Uncontrolled illness including, but not limited to, ongoing or active infection (other than chronic viral infections that are controlled, e.g. HIV, as described above), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (uncontrolled), cirrhosis, or psychiatric illness/ social situations that would limit compliance with the study requirements.
* Patients with prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Indwelling catheters (e.g., PleurX®) are allowed.
* Corrected serum Ca > 12 mg/dl.
* Patients who are receiving hypocalcemic therapies (e.g. denosumab, bisphosphonates) who achieve appropriate serum calcium levels are eligible.
* Pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 6 years
  To estimate the ORR including confirmed complete response (CR) and partial response (PR) rates in each treatment group 1-3

SECONDARY OUTCOMES:
Frequency of adverse events | 6 years
  To evaluate the frequency and severity of toxicities attributed to chemotherapy administered on trial. To evaluate the tolerability of prospectively dose attenuated chemotherapy
  Evaluate toxicity by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 5.0 criteria (CTCAE 5.0) by Treatment Group in all patients who received at least one dose of treatment on trial.
  Tolerability will be defined as receiving two or more chemotherapy cycles with no more than a one week delay (due to treatment related toxicity) during the initial treatment period (first four cycles), delivered with pre-specified dose modifications to the cytotoxic component(s) of standard regimens for NSCLC and SCLC. Proportions of adverse events will be tabulated and organized by grade (all grade and grade 3 or higher).
Progression free survival (PFS) | 6 years
  To evaluate PFS in each treatment group. PFS is defined as the time from treatment initiation until documented disease progression, clinical progression, death, or the end of follow-up, whichever occurs first. Patients who are still alive and progression free at last follow-up will be considered censored at the time of last tumor assessment
Overall survival (OS) | 6 years
  To evaluate overall survival (OS) in each treatment group. OS is defined as the time from treatment initiation until death. Patients who are still alive at end of follow-up will be considered censored.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Judd, DO, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No